CLINICAL TRIAL: NCT03876132
Title: Multifactorial Analysis of the Influence of Alcohol Marketing Stimuli Among Young Adults on the Perception of the Risks of Alcohol and According to the Types of Uses and Individual Vulnerabilities
Brief Title: Perception of the Risks of Alcohol and Individual Vulnerabilities in Young Adults
Acronym: DEPREV
Status: Terminated | Type: Observational
Why Stopped: The number of patients is suffisant to answer to the primary outcome
Sponsor: University Hospital, Brest (Other)
Collaborators: Ecole des Hautes Etudes en Santé Publique (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC19.0059_DEPREV
Record Dates: First submitted 2019-03-11; First posted 2019-03-15 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Alcohol Abuse
Keywords: regular consumption of alcohol; young adults; Moderate or severe alcohol use disorders
MeSH Terms: conditions — Alcoholism; Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Alcohol use is the second leading cause of preventable death after smoking. The Evin law was built in 1991 with the goal of reducing exposure to alcohol marketing among the youngest. But this law is currently extremely weakened, and in a press release of February 26, 2018, the French Society of Alcoology is alarmed by these developments.

Studies focusing on the impact of alcohol marketing focus largely on young adolescents, and the links between exposure to marketing and the initiation of alcohol. But beyond these links, there has been little work on the impact of alcohol marketing in vulnerable subjects with regular alcohol consumption. Consumption of alcohol is one of the first causes of hospitalization in France (Paille and Reynaud, 2015), the damage is often restricted to notions of dependency risks, but they can appear as soon as consumptions of 1 US / d (Guerin and Laplanche, 2013) and they mainly concern 45-64 year olds. To our knowledge, there are no studies on the impact of alcohol marketing conducted on regular alcohol users, depending on how they use alcohol (use, or use disorders). mild, moderate or severe) in patients enrolled in primary care and specialized addiction care.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 45 years with moderate or severe alcohol use disorders
* Followed in addiction at Brest CHRU

Exclusion Criteria:

* Major from 18 to 45 years
* Current consumption of alcohol (multi-monthly)
* Follow-up in primary care or addictology in Brest

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients aged 18 to 45 years, followed in addictology or hospitalized in addictology at the Brest University Hospital with moderate or severe alcohol use disorders Major subjects (18-45 years) followed in primary care, meeting the inclusion criteria, with a selection according to level of disorder of alcohol use (absence, mild or moderate disorders). The interview will be integrated into the care in primary care.
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2019-11-14 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Alcohol craving | 1 day
  Evaluation of alcohol craving, evaluated by a visual analogue scale from 0 to 100. It is in the form of a straight line of 100 mm. In one ends is indicated: absence of pain, to the other: unbearable pain. The patient places a marks between these two ends depending on the intensity of his pain at a given time. In practice, it is a small plastic strip provided, on a face of a cursor mobilized by the patient, on the other with millimeter graduations read by the caregiver.

SECONDARY OUTCOMES:
Level of anxiety | 1 day
  Assessment of the level of anxiety felt before and after the interview evaluated by a visual analogue scale from 0 to 100
Perceived risks | 1 day
  Evaluation of perceived risks related to stimuli by individual interviews following the presentation of advertising images. It is not a scale but in interview where feelings are raised. No score.
Sensitivity to stimuli | 1 day
  Assessment of sensitivity to stimuli presented
Attractiveness of stimuli | 1 day
  Evaluation of the attractiveness of stimuli by individual interviews following the presentation of advertising images. It is not a scale but in interview where feelings are raised. No score.
Alcohol consumed | 1 day
  Evaluation of the categories of alcohol consumed

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning five years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement

REFERENCES:
- [Derived] Guillou-Landreat M, Dany A, Le Reste JY, Le Goff D, Benyamina A, Grall-Bronnec M, Gallopel-Morvan K. Impact of alcohol marketing on drinkers with Alcohol use disorders seeking treatment: a mixed-method study protocol. BMC Public Health. 2020 Apr 7;20(1):467. doi: 10.1186/s12889-020-08543-6. PMID 32264848